CLINICAL TRIAL: NCT06040294
Title: Evaluation of a Dementia and Disability Simulation Program for Senior Activity Facilitation Skills Among College Nursing Students
Brief Title: Dementia and Disability Simulation for College Nursing Students' Senior Activity Facilitation Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tzu Chi University (Other)
Responsible Party: Principal Investigator, Huei-Chuan Sung, Associate professor, Tzu Chi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: YLH-IRB-11210
Record Dates: First submitted 2023-09-09; First posted 2023-09-15 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Dementia
Keywords: dementia; disability; simulation; nursing student
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: two-group randomised controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dementia and disability simulation program (DDS) (Experimental): DDS program consists of dementia virtual reality and disability simulation of activity design for seniors
  Interventions: Other: DDS program
- dementia course with no DDS (Active Comparator): Regular dementia course and group discussions of activity design for seniors with no DDS
  Interventions: Other: dementia course with no DDS

INTERVENTIONS:
Other: DDS program — dementia virtual reality and disability simulation of activity design for seniors
  Arms: dementia and disability simulation program (DDS)
Other: dementia course with no DDS — Regular dementia course and group discussions of activity design for seniors with no DDS
  Arms: dementia course with no DDS

SUMMARY:
This study aims to evaluate the effectiveness of a dementia and disability simulation (DDS) program on dementia knowledge, attitude, empathy, and activity design skills for seniors among college nursing students.

DETAILED DESCRIPTION:
This two-group randomised controlled trial aims to evaluate the effectiveness of a dementia and disability simulation program on dementia knowledge, attitude, empathy, and activity design skills for seniors among college nursing students.

The interventional group will receive a 6-week dementia and disability simulation program of activity design for seniors.

The control group will receive 6 weeks of regular dementia course and group discussion of activity design for seniors with no dementia and disability simulation.

Both groups will be assessed for their dementia knowledge, attitude, empathy and activity design skills for seniors at baseline, week 12, and week 18.

ELIGIBILITY:
Inclusion Criteria:

* college nursing students with age ranged from 19 to 40 years,
* Taiwanese nationality,
* Sophomore and above
* provide informed consent to participate in the study.

Exclusion Criteria:

-college nursing students who do not meet the inclusion criteria

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-09-07 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Dementia Knowledge Assessment Scale (DKAS) | Baseline, week 12, week 18
  score of knowledge about dementia (0~50) higher scores indicate more knowledge about dementia
Approaches to Dementia Questionnaire (ADQ) | Baseline, week 12, week 18
  score of attitude toward people with dementia (19~95) higher scores indicate more positive attitude towards dementia
Jefferson Scale of Empathy (JSE) | Baseline, week 12, week 18
  score of empathy (20~140) higher scores indicate more empathy for people with dementia
Rubrics of activity design skills for seniors | Baseline, week 12, week 18
  score of activity design skills for seniors (0~45) higher scores indicate better skills of designing activities for seniors

CONTACTS AND LOCATIONS:
Overall Officials: Huei-Chuan Sung, PhD, Principal Investigator — Tzu Chi University
Locations (1):
- Tzu Chi University, Hualien City, Taiwan